CLINICAL TRIAL: NCT00385983
Title: Total Thyroidectomy With Harmonic Scalpel® Versus Standard Surgery. Open Multicentric Randomized Controlled Trial
Brief Title: Total Thyroidectomy With Harmonic Scalpel®
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brazilian Society of Head and Neck Surgery (Other)
Collaborators: Johnson & Johnson (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP005
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Thyroid Neoplasm; Goiter; Thyroid Nodule
Keywords: thyroidectomy; thyroid neoplasm; postoperative complications; cost effectiveness
MeSH Terms: conditions — Thyroid Neoplasms; Goiter; Thyroid Nodule; Postoperative Complications

INTERVENTIONS:
Device: Harmonic Scalpel

SUMMARY:
Harmonic scalpel is a new surgical instrument. Its use has been recommended in patients submitted to total thyroidectomy. Few randomized controlled trials has been published. However they had small sample sizes, used intermediate outcomes and included different surgical procedures.

Our objective is to asses the use of Harmonic scalpel in patients submitted to total thyroidectomy using surgical complications, operative time, drainage volume, postoperative pain, length of stay and costs as outcomes. Our hypothesis is that Harmonic scalpel decreases operative time,drainage volume, postoperative pain, length of stay and costs without increasing surgical complications

DETAILED DESCRIPTION:
This is a multicentric open phase IV randomized controlled trial comparing patients submitted to total thyroidectomy comparing standard surgical procedure versus Harmonic scalpel assisted procedure. Adult patients with benign or malignant thyroid disease and normal function will be included. Patients with giant goiter, hyperthyroidism, non differentiated thyroid carcinoma, locally invasive tumors, neck dissection, previous neck radiotherapy or chemotherapy, video assisted surgery and severe comorbidities will be excluded. calculated sample size was 280 patients. Outcomes will be assessed by an independent monitor. All centers will made a previous standardization of surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 y/o)
* Benign or malignant thyroid disease
* Proposal of total thyroidectomy
* Normal thyroid function

Exclusion Criteria:

* Giant goiter
* Hyperthyroidism
* Non differentiated thyroid carcinoma
* Locally invasive tumors
* Neck dissection as a part of procedure
* Previous surgery, radiotherapy or I131 therapy on neck
* Video-assisted or endoscopic thyroidectomy
* Severe comorbidities
* Coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280

PRIMARY OUTCOMES:
Postoperative complications

SECONDARY OUTCOMES:
Operative time
Drainage volume
Postoperative pain
Length of stay
Direct Costs

CONTACTS AND LOCATIONS:
Overall Officials: Luiz P Kowalski, PhD, Principal Investigator — Brazilian Society of Head and Neck Surgery
Locations (9):
- Brazil (9):
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Instituto Nacional de Cancer INCA, Rio de Janeiro, Rio de Janeiro
  - Hospital do Cancer de Natal, Natal, Rio Grande do Norte
  - Hospital do Cancer AC Camargo, São Paulo, São Paulo
  - Hospital Heliopolis, São Paulo, São Paulo
  - Hospital Sao Paulo-UNIFESP, São Paulo, São Paulo
  - Instituto Arnaldo Vieira de Carvalho, São Paulo, São Paulo
  - Santa Casa de Misericordia, São Paulo, São Paulo